CLINICAL TRIAL: NCT05671809
Title: Effects of Different Treatment for Anorectal Function of Patients With Rectal Cancer: a Study Protocol for a Prospective, Observational, Controlled, Multicentre Study
Brief Title: Effects of Different Treatment for Anorectal Function of Patients With Rectal Cancer
Acronym: ARF-RC
Status: Not yet recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-097
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-11

CONDITIONS: Rectal Cancer
Keywords: Anorectal function, Rectal cancer, NCRT, Surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NCRT with surgery: Rectal cancer patients who will undergo sphincter-preserving therapy, that is NCRT with surgery.
  Interventions: Other: NCRT with surgery, or NCT with surgery, or surgery
- NCT with surgery: Rectal cancer patients who will undergo sphincter-preserving therapy, that is NCT with surgery.
  Interventions: Other: NCRT with surgery, or NCT with surgery, or surgery
- surgery: Rectal cancer patients who will undergo sphincter-preserving therapy, that is surgery.
  Interventions: Other: NCRT with surgery, or NCT with surgery, or surgery

INTERVENTIONS:
Other: NCRT with surgery, or NCT with surgery, or surgery — The eligible patients who voluntarily sign the consent form will undergo either NCRT with surgery, or NCT with surgery, or surgery according to treatment guidelines.

SUMMARY:
Background

Neoadjuvant chemoradiotherapy (NCRT) and total mesorectal excision are standard treatments for patients with locally advanced rectal cancer. These sphincter-saving operations may be accompanied by a series of functional disorders. Prospective studies dynamically evaluating the different roles of surgery and NCRT on anorectal function are lacking.

Methods/design

The study is a prospective, observational, controlled, multicentre study. After screening for eligibility and obtaining informed consent, a total of 402 rectal cancer patients aged from 18 to 75 years old undergoing sphincter preservation treatments at The Sixth Affiliated Hospital, Sun Yat-sen University and Nanfang Hospital, Southern Medical University are included in the trial. The primary outcome measure is the average resting pressure of anal sphincter. The secondary outcome measures are maximum anal sphincter contraction pressure and Wexner continence score. Evaluations will be carried out at the following stages: baseline (T1), after radiotherapy or chemotherapy (before surgery, T2), after surgery (before closing the temporary stoma, T3), and at follow-up visits (every 3 to 6 months, T4, T5……). Follow-up for each patient will be at least 2 years.

Discussion

We expect the program to provide more information on therapeutical options and strategies to reduce anorectal dysfunction of rectal cancer patients who have been undergone sphincter preservation treatments.

DETAILED DESCRIPTION:
Study design and setting

The study is a prospective, observational, controlled, multicentre study of patients diagnosed with rectal cancer. The eligible patients will be informed about the study in detail. After providing written informed consent, these patients will undergo sphincter-preserving therapies including either NCRT with surgery, or NCT with surgery or surgery. All patients will receive anorectal manometry and Wexner continence score before and after therapies and at follow-up visits.

Participants

Patients diagnosed with rectal cancer at The Sixth Affiliated Hospital, Sun Yat-sen University and Nanfang Hospital, Southern Medical University will be assessed for suitability for inclusion.

Inclusion criteria

18-75 years of age. Rectal cancer with pathological diagnosis. Patient will undergo sphincter-preserving therapies. ECOG score for performance status is 0-2. Written informed consent.

Exclusion criteria

Patients who have undergone rectal cancer surgery. Patients who have received pelvic radiotherapy. Patients with other active malignant tumors. Recently (less than 4 weeks) received surgery or patients with recent severe trauma.

Significant cardiac disease: congestive heart failure of New York Heart Association class ≥2; patients with recent (less than 12 months) active coronary artery disease (unstable angina or myocardial infarction).

Recent (less than 6 months) thrombosis or embolism events, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism and deep vein thrombosis.

Patients with toxicity (CTCAE Grade ≥ 2) caused by previous treatment that has not subsided.

Pregnant or lactating women.

Interventions

The eligible patients who voluntarily sign the consent form will undergo either NCRT with surgery, or NCT with surgery, or surgery according to treatment guidelines.

Outcomes

Evaluations will take place at baseline (T1), after radiotherapy or chemotherapy (before surgery, T2), after surgery (before closing the temporary stoma, T3), and at follow-up visits (every 3 to 6 months, T4, T5……). Follow-up for each patient will be at least 2 years.

The primary outcome is the average resting pressure (ARP) of anal sphincter. The secondary outcomes are maximum anal sphincter contraction pressure and Wexner continence score. High-resolution anorectal manometry will be used to assess the average resting pressure and maximal contraction pressure. We will use high-resolution anorectal manometry with a 24-channel water-perfused catheter (Multiplex, Alacer, Biomedica, Sao Paulo, Brazil), which has proven to be adequate for clinical use. This test will be performed by a trained physician. In addition, we will use Wexner continence score to assess fecal incontinence symptoms and their impact on the quality of life of patients following sphincter-preserving rectal cancer surgery.

Recruitment

Patients aged 18-75 years who have been diagnosed with rectal cancer and consider sphincter-preserving therapies are eligible for the study. The study physicians will inform the patients about the study in detail. After obtaining informed consent, the patient is recruited to the study.

Allocation

The study is a prospective, observational, controlled study without randomization. Treatment decisions will be made by multidisciplinary team for eligible patients who voluntarily sign the consent form. All patients will receive evaluation of the anorectal function through anorectal manometry and Wexner continence score before and after therapies and at follow-up visits.

Participant timeline

Recruitment started in December 2022 at The Sixth Affiliated Hospital, Sun Yat-sen University and Nanfang Hospital, Southern Medical University.

Sample size

The sample size calculation was performed considering the results of a previous case-control study with rectal cancer patients undergoing chemoradiotherapy and/or surgery. In this study, RP was significantly lower in the chemoradiotherapy group than in the surgery group (32.7 +/- 17 vs 45.3 +/- 18 mmHg; P =.03) at the time of ileostomy closure. These values were introduced at PASS v11 software (NCSS, LLC. Kaysville, Utah, USA) with a power of 80%, alpha 0.05, and an enrollment ratio of 1/1, resulting in an estimated sample size of 122 participants in each group. Then, considering the need of lost to follow-up, which is estimated at around 10.0% of the cases, we will require a total of 134 patients in each group.

Data management, collection and monitoring

All protocol-required information collected during the study will be entered by the investigator in the electronic case report forms (CRF). The investigator should complete the CRF as soon as possible after information is collected. An explanation should be given for all missing data. The completed CRF will be reviewed and signed by the investigator. The main investigator will continuously monitor data. Data will be stored in the secured network of Sun Yat-sen University and for security reasons, in an external hard drive which will be used to back up regularly the database.

Statistical methods

For statistical analysis of the quantitative variables with normal distribution, the mean, standard deviation (SD), median and interquartile range will be calculated. Group comparisons will be made using t tests or Mann-Whitney U test for continuous variables. Associations between the categorical variables will be tested with the Chi-Square-test or the Fisher exact test, when appropriate. Paired values (before and after therapies) will be compared for each patient using a paired t test or a Wilcoxon test. The data will be analyzed using IBM SPSS Statistics for Windows, version 27.0 (IBM Corporation, Armonk, NY, USA). A significance threshold of p < 0.05 will be adopted for all tests.

Research ethic approval

The study adheres to the Declaration of Helsinki on medical research protocols and ethics. The protocol was reviewed and approved by the Human Medical Ethics Committee of the Sixth Affiliated Hospital of Sun Yat-sen University (number 2022ZSLYEC-614).

ELIGIBILITY:
Inclusion Criteria:

18-75 years of age. Rectal cancer with pathological diagnosis. Patient will undergo sphincter-preserving therapies. ECOG score for performance status is 0-2. Written informed consent.

Exclusion Criteria:

Patients who have undergone rectal cancer surgery. Patients who have received pelvic radiotherapy. Patients with other active malignant tumors. Recently (less than 4 weeks) received surgery or patients with recent severe trauma.

Significant cardiac disease: congestive heart failure of New York Heart Association class ≥2; patients with recent (less than 12 months) active coronary artery disease (unstable angina or myocardial infarction).

Recent (less than 6 months) thrombosis or embolism events, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism and deep vein thrombosis.

Patients with toxicity (CTCAE Grade ≥ 2) caused by previous treatment that has not subsided.

Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with rectal cancer at The Sixth Affiliated Hospital, Sun Yat-sen University and Nanfang Hospital, Southern Medical University will be assessed for suitability for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ARP | Baseline (T1), after radiotherapy or chemotherapy (before surgery, T2), after surgery (before closing the temporary stoma, T3), follow-up visits (every 3 to 6 months, T4, T5……)
  The average resting pressure (ARP) of anal sphincter

SECONDARY OUTCOMES:
MASCP and Wexner | Baseline (T1), after radiotherapy or chemotherapy (before surgery, T2), after surgery (before closing the temporary stoma, T3), follow-up visits (every 3 to 6 months, T4, T5……)
  Maximum anal sphincter contraction pressure and Wexner continence score

CONTACTS AND LOCATIONS:
Overall Officials: Xin-juan Fan, Ph.D, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University; Xiang-Bo Wan, Ph.D, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University; Hong-Cheng Lin, Ph.D, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Newland RC, Chapuis PH, Dent OF, Bokey EL. Total mesorectal excision is optimal surgery for rectal cancer: a Scandinavian consensus. Br J Surg. 1996 Mar;83(3):427-8. doi: 10.1002/bjs.1800830355. No abstract available. PMID 8665225
- [Background] Keller DS, Berho M, Perez RO, Wexner SD, Chand M. The multidisciplinary management of rectal cancer. Nat Rev Gastroenterol Hepatol. 2020 Jul;17(7):414-429. doi: 10.1038/s41575-020-0275-y. Epub 2020 Mar 12. PMID 32203400
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Sauer R, Liersch T, Merkel S, Fietkau R, Hohenberger W, Hess C, Becker H, Raab HR, Villanueva MT, Witzigmann H, Wittekind C, Beissbarth T, Rodel C. Preoperative versus postoperative chemoradiotherapy for locally advanced rectal cancer: results of the German CAO/ARO/AIO-94 randomized phase III trial after a median follow-up of 11 years. J Clin Oncol. 2012 Jun 1;30(16):1926-33. doi: 10.1200/JCO.2011.40.1836. Epub 2012 Apr 23. PMID 22529255
- [Background] Sipaviciute A, Sileika E, Burneckis A, Dulskas A. Late gastrointestinal toxicity after radiotherapy for rectal cancer: a systematic review. Int J Colorectal Dis. 2020 Jun;35(6):977-983. doi: 10.1007/s00384-020-03595-x. Epub 2020 Apr 16. PMID 32296933
- [Background] Bryant CL, Lunniss PJ, Knowles CH, Thaha MA, Chan CL. Anterior resection syndrome. Lancet Oncol. 2012 Sep;13(9):e403-8. doi: 10.1016/S1470-2045(12)70236-X. PMID 22935240
- [Background] Celerier B, Denost Q, Van Geluwe B, Pontallier A, Rullier E. The risk of definitive stoma formation at 10 years after low and ultralow anterior resection for rectal cancer. Colorectal Dis. 2016 Jan;18(1):59-66. doi: 10.1111/codi.13124. PMID 26391723
- [Background] De Nardi P, Testoni SG, Corsetti M, Andreoletti H, Giollo P, Passaretti S, Testoni PA. Manometric evaluation of anorectal function in patients treated with neoadjuvant chemoradiotherapy and total mesorectal excision for rectal cancer. Dig Liver Dis. 2017 Jan;49(1):91-97. doi: 10.1016/j.dld.2016.09.005. Epub 2016 Sep 22. PMID 27720700
- [Background] Sun W, Dou R, Chen J, Lai S, Zhang C, Ruan L, Kang L, Deng Y, Lan P, Wang L, Wang J. Impact of Long-Course Neoadjuvant Radiation on Postoperative Low Anterior Resection Syndrome and Quality of Life in Rectal Cancer: Post Hoc Analysis of a Randomized Controlled Trial. Ann Surg Oncol. 2019 Mar;26(3):746-755. doi: 10.1245/s10434-018-07096-8. Epub 2018 Dec 7. PMID 30536129
- [Background] Bharucha AE. Update of tests of colon and rectal structure and function. J Clin Gastroenterol. 2006 Feb;40(2):96-103. doi: 10.1097/01.mcg.0000196190.42296.a9. PMID 16394868
- [Background] Kitaguchi D, Nishizawa Y, Sasaki T, Tsukada Y, Ito M. Clinical benefit of high resolution anorectal manometry for the evaluation of anal function after intersphincteric resection. Colorectal Dis. 2019 Mar;21(3):335-341. doi: 10.1111/codi.14528. Epub 2018 Dec 31. PMID 30537066
- [Background] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Background] Chen SC, Futaba K, Leung WW, Wong C, Mak T, Ng S, Gregersen H. Functional anorectal studies in patients with low anterior resection syndrome. Neurogastroenterol Motil. 2022 Mar;34(3):e14208. doi: 10.1111/nmo.14208. Epub 2021 Jun 18. PMID 34145694
- [Background] Birnbaum EH, Dreznik Z, Myerson RJ, Lacey DL, Fry RD, Kodner IJ, Fleshman JW. Early effect of external beam radiation therapy on the anal sphincter: a study using anal manometry and transrectal ultrasound. Dis Colon Rectum. 1992 Aug;35(8):757-61. doi: 10.1007/BF02050325. PMID 1643999
- [Background] Lim JF, Tjandra JJ, Hiscock R, Chao MW, Gibbs P. Preoperative chemoradiation for rectal cancer causes prolonged pudendal nerve terminal motor latency. Dis Colon Rectum. 2006 Jan;49(1):12-9. doi: 10.1007/s10350-005-0221-7. PMID 16292664
- [Background] Bjoern MX, Perdawood SK. Manometric assessment of anorectal function after transanal total mesorectal excision. Tech Coloproctol. 2020 Mar;24(3):231-236. doi: 10.1007/s10151-020-02147-3. Epub 2020 Feb 1. PMID 32008213
- [Background] Fratta CL, Pinheiro LV, Costa FO, Magro DO, Martinez CAR, Coy CSR. STUDY OF ANORECTAL PHYSIOLOGY PRE AND POS NEOADJUVANT THERAPY FOR RECTAL CANCER BY ANORECTAL MANOMETRY AND JORGE-WEXNER SCORE. Arq Gastroenterol. 2022 Jul-Sep;59(3):334-339. doi: 10.1590/S0004-2803.202203000-61. PMID 36102428
- [Background] Ammann K, Kirchmayr W, Klaus A, Muhlmann G, Kafka R, Oberwalder M, De Vries A, Ofner D, Weiss H. Impact of neoadjuvant chemoradiation on anal sphincter function in patients with carcinoma of the midrectum and low rectum. Arch Surg. 2003 Mar;138(3):257-61. doi: 10.1001/archsurg.138.3.257. PMID 12611569
- [Derived] Shi J, Cheng YK, He F, Zheng J, Wang YL, Wan XB, Lin HC, Fan XJ. Effects of neoadjuvant radiochemotherapy for anorectal function in locally advanced rectal cancer patients: a study protocol for a prospective, observational, controlled, multicentre study. BMC Cancer. 2023 May 22;23(1):467. doi: 10.1186/s12885-023-10951-x. PMID 37217903